CLINICAL TRIAL: NCT02288832
Title: Medico-economic Impact of Screening Atopobium Vaginae and Gardnerella Vaginalis in Molecular Biology by "Point-of-care" During Pregnancy
Acronym: AuTop
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2014-001559-22; RCAPHM14_0085 (Other: AP HM)
Record Dates: First submitted 2014-10-30; First posted 2014-11-11 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2015-11

CONDITIONS: Low Risk of Preterm Delivery
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Innovative strategy (group A): (Experimental): these women will undergo routine screening for bacterial vaginosis by analysis of their self-collected vaginal samples with this innovative technique; if the test is found to be positive, an appropriate treatment will be prescribed. The POC (point-of-care) test will be considered positive if: A. vaginae is detected at a threshold > 105.copies per ml and/or G. vaginalis > 105 copies per ml. The women with vaginosis will be screened monthly for recurrences through 28 weeks, and recurrence will be treated.
  Interventions: Other: -self-collected vaginal samples; Drug: zithromax
- Standard strategy (group B): (Other): This group will be followed according to the usual practices of the physicians seeing them.
  Interventions: Other: usual practices

INTERVENTIONS:
Other: -self-collected vaginal samples
  Arms: Innovative strategy (group A):
Drug: zithromax
  Other Names: azithromycine
  Arms: Innovative strategy (group A):
Other: usual practices
  Arms: Standard strategy (group B):

SUMMARY:
Infection is the principal cause of preterm births. Most (90%) women with preterm deliveries have no abnormal history. It is widely agreed that preterm delivery is often associated with bacterial vaginosis. One of the major difficulties at this time is that the diagnosis of bacterial vaginosis is based on heterogeneous criteria. The technique currently used is the Nugent score, but it lacks the characteristics necessary for widespread use in the general population. It must be performed on a fresh swab, and any delay in transporting it can cause drying that makes the test difficult to perform.

The investigators have developed a rapid diagnostic tool for bacterial vaginosis using molecular biology based on a point of care model and obtained a patent (European Patent Office N° 2087134). In comparison with the reference techniques, our tool's performance has been excellent, in terms of specificity, sensitivity, and positive and negative predictive values. In particular, our work showed that 57% of the flora samples rated as intermediate on the Nugent score were in reality true bacterial vaginosis. Molecular biology therefore identifies a homogeneous population of women with vaginal flora anomalies. The investigators recently showed that the carriage of Atopobium vaginae and/or Gardnerella vaginalis >105/mL shortens the time to delivery in a population at risk of preterm delivery (PHRC 2006). Vaginal flora anomalies are therefore an important target for preventing preterm delivery.

DETAILED DESCRIPTION:
The principal objective is to use a cost-effectiveness study to assess the medical and economic impact of a new strategy for the screening and subsequent treatment of vaginal flora anomalies before the 20th week of gestation- molecular biology techniques (PCR for A. vaginae and G. vaginalis by point-of-care testing) will test self-collected vaginal samples in a population of pregnant women at low risk of preterm delivery. There are multiple secondary objectives, including assessment of the effect of the strategy on the following indicators- delivery before 26, 32, and 37 weeks. Methods-An open-label prospective randomized study will compare 2 groups with different management of their pregnancies. Pregnant women at low risk, regardless of any symptoms, will be randomized into 2 groups. The study will not include women at high risk of preterm delivery. Innovative strategy (group A)- these women will undergo routine screening for bacterial vaginosis by analysis of their self-collected vaginal samples with this innovative technique.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years with a pregnancy before 20 weeks are some parity and gravidity;
* Woman who understood the process and the objectives of the study and who agreed to sign an informed consent;
* Without a history of premature birth or late abortion (population at low risk of preterm birth);
* Having no major risk factors for prematurity: insulin-dependent diabetes, systemic lupus erythematosus, hypertension, uterine malformation, cone biopsy, multiple pregnancy;
* No pre-existing hypertension;
* Asymptomatic or symptomatic regarding the diagnosis of bacterial vaginosis.

Exclusion Criteria:

* Woman withdrawing her consent during the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6800 (Actual)
Dates: Start 2015-03-06 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
the incremental cost-effectiveness | 30 months
  the incremental cost-effectiveness ratio between the two groups corresponding to the cost of preterm birth before 37 avoided.
  * average differential effect in terms of preterm birth before 37 weeks of 0.013. A preterm birth rate of 0.043 (+/- 0.043) is expected in the group B and 0.03 (+/- 0.03) in Group A;
  * Cost differential means € 230 +/- 35. This difference takes into account the estimated EFC (initial and recurrent) cost and estimated cost of treatments vaginosis cases (10% of patients);
  * Cost-effectiveness threshold of 22,500 euros corresponding to the average cost ratio that is could avoid caring for a child born prematurely before 37 weeks as documented in the international literature (Petrou 2012);

SECONDARY OUTCOMES:
the delivery rate before 26, 28, 32 and 37 weeks | 30 months
the rate of rupture of membranes | 30 months
the rate of intrauterine growth retardation | 30 months
the rate of endometritis | 30 months
the preterm birth rate adjusted | 30 months
he total duration of hospitalization and earlier for postpartum mother and newborn in number of days | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle DESALBRES, Study Director — Assistance Publique Hopitaux De Marseille
Locations (2):
- France (2):
  - Assistance Publique Hopitaux de Marseille, Marseille
  - Hôpital Nord Assistance Publique Hôpitaux de Marseille, Marseille

REFERENCES:
- [Derived] Bretelle F, Loubiere S, Desbriere R, Loundou A, Blanc J, Heckenroth H, Schmitz T, Benachi A, Haddad B, Mauviel F, Danoy X, Mares P, Chenni N, Menard JP, Cocallemen JF, Slim N, Senat MV, Chauleur C, Bohec C, Kayem G, Trastour C, Bongain A, Rozenberg P, Serazin V, Fenollar F; Groupe de Recherche en Obstetrique et Gynecologie (GROG) Investigators. Effectiveness and Costs of Molecular Screening and Treatment for Bacterial Vaginosis to Prevent Preterm Birth: The AuTop Randomized Clinical Trial. JAMA Pediatr. 2023 Sep 1;177(9):894-902. doi: 10.1001/jamapediatrics.2023.2250. PMID 37459059
- [Derived] Bretelle F, Fenollar F, Baumstarck K, Fortanier C, Cocallemen JF, Serazin V, Raoult D, Auquier P, Loubiere S. Screen-and-treat program by point-of-care of Atopobium vaginae and Gardnerella vaginalis in preventing preterm birth (AuTop trial): study protocol for a randomized controlled trial. Trials. 2015 Oct 19;16:470. doi: 10.1186/s13063-015-1000-y. PMID 26482128